CLINICAL TRIAL: NCT04295551
Title: Multicenter Clinical Study on the Efficacy and Safety of Xiyanping Injection in the Treatment of New Coronavirus Infection Pneumonia (General and Severe)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QF-XYP1990-1
Record Dates: First submitted 2020-03-03; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group of ordinary COVID-19 (Experimental): Lopinavir / ritonavir tablets combined with Xiyanping injection
  Interventions: Drug: Lopinavir / ritonavir tablets combined with Xiyanping injection
- Control group of ordinary COVID-19 (Active Comparator): ritonavir/ritonavir treatment
  Interventions: Drug: Lopinavir/ritonavir treatment
- Experimental group of severe COVID-19 (Experimental): Lopinavir / ritonavir tablets combined with Xiyanping injection
  Interventions: Drug: Lopinavir / ritonavir tablets combined with Xiyanping injection

INTERVENTIONS:
Drug: Lopinavir / ritonavir tablets combined with Xiyanping injection — Xiyanping injection, 10-20ml daily, Qd, the maximum daily does not exceed 500mg (20mL) + Lopinavir tablet or Ritonavir tablet+Alpha-interferon nebulization, for 7-14 days,
  Arms: Experimental group of ordinary COVID-19; Experimental group of severe COVID-19
Drug: Lopinavir/ritonavir treatment — Lopinavir / ritonavir tablets, 2 times a day, 2 tablets at a time; alpha-interferon nebulization
  Arms: Control group of ordinary COVID-19

SUMMARY:
In December 2019, Wuhan, in Hubei province, China, became the center of an outbreak of pneumonia of unknown cause. In a short time, Chinese scientists had shared the genome information of a novel coronavirus (2019-nCoV) from these pneumonia patients and developed a real-time reverse transcription PCR (real time RT-PCR) diagnostic assay.

In view of the fact that there is currently no effective antiviral therapy, the prevention or treatment of lung injury caused by COVID-19 can be an alternative target for current treatment. Xiyanping injection has anti-inflammatory and immune regulation effects. This study is a Randomized, Parallel Controlled Clinical Study to treat patients with COVID-19 infection.

DETAILED DESCRIPTION:
The new coronavirus (COVID-19) [1] belongs to the new beta coronavirus. Current research shows that it has 85% homology with bat SARS-like coronavirus (bat-SL-CoVZC45), but its genetic characteristics are similar to SARSr-CoV. There is a clear difference from MERSr-COV. Since December 2019, Wuhan City, Hubei Province has successively found multiple cases of patients with pneumonia infected by a new type of coronavirus. With the spread of the epidemic, as of 12:00 on February 12, 2020, a total of 44726 confirmed cases nationwide (Hubei Province) 33,366 cases, accounting for 74.6%), with 1,114 deaths (1068 cases in Hubei Province), and a mortality rate of 2.49% (3.20% in Hubei Province).

In view of the fact that there is currently no effective antiviral therapy, the prevention or treatment of lung injury caused by COVID-19 can be an alternative target for current treatment. Xiyanping injection has anti-inflammatory and immune regulation effects. In the early clinical practice of treating severe H1N1, it was clinically concerned, and combined with conventional treatment, and achieved good results.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >=18 years;
2. Novel coronavirus pneumonia patients diagnosed by pathogenic testing;
3. The patient himself participated in the study voluntarily, agreed and signed the informed consent.

Exclusion Criteria:

1. Meet the diagnostic criteria for severe new-type coronavirus infection pneumonia;
2. Severe primary diseases that affect survival, including: uncontrolled malignant tumors, hematological diseases, and HIV that have not been metastasized in multiple places;
3. Obstructive pneumonia, pulmonary interstitial fibrosis, alveolar proteinosis, and allergic alveolitis caused by lung tumors;
4. Women who are breastfeeding or pregnant;
5. Those who are known to be allergic to the ingredients contained in the research medication, or patients with allergies;
6. Those who have continued to use immunosuppressive agents or organ transplants in the past 6 months;
7. Patients who have participated in other drug clinical trials within 3 months before the screening test;
8. The investigator judges that he or she cannot complete or should not participate in the study (expected death within 48 hours, and the patient refuses active treatment)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-14 (Estimated); Primary Completion 2020-07-14 (Estimated); Study Completion 2021-04-14 (Estimated)

PRIMARY OUTCOMES:
Clinical recovery time | Up to Day 28
  The time from study drug use to complete fever reduction and cough recovery is measured in hours.